CLINICAL TRIAL: NCT05529628
Title: The Cytokines and Immune Checkpoint Differences Between Fournier Gangrene and Perianal Abscess
Brief Title: The Immunological Differences Between Fournier Gangrene and Perianal Abscess
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD. PhD, Istanbul Training and Research Hospital
Other Study IDs: Fournier Gangrene
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Fournier Gangrene; Perianal Abscess
Keywords: Cytokine; inflammation; Fournier Gangrene; Perianal Abscess
MeSH Terms: conditions — Fournier Gangrene; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Healthy volunteers with no known chronic or cancer disease
  Interventions: Diagnostic Test: Cytokine levels
- Fournier's gangrene: Fournier's gangrene patients
  Interventions: Diagnostic Test: Cytokine levels
- Perianal abscess: Perianal abscess patients
  Interventions: Diagnostic Test: Cytokine levels

INTERVENTIONS:
Diagnostic Test: Cytokine levels — Preoperative cytokine levels of the patients

SUMMARY:
Although it is rarely observed, necrotizing fasciitis progresses with high mortality and serious complications. Fournier's gangrene is a specific form of necrotizing fasciitis. In laboratory tests, leukocytosis or leukopenia, anemia, lymphopenia can be observed. Perianal abscess is a surgical emergency that is observed much more frequently than necrotizing fasciitis. Although Fournier's gangrene has many different etiologies, it rarely occurs due to the progression of perianal abscess, and although it is difficult to distinguish between these two diseases at diagnosis, the two diseases manifest themselves as different entities. In this study, blood cytokine levels will be evaluated in patients with Fournier's gangrene and perianal abscess, and the role of blood cytokine levels in the differential diagnosis of these two diseases will be investigated.

DETAILED DESCRIPTION:
Although it is rarely observed, necrotizing fasciitis progresses with high mortality and serious complications. Fournier's gangrene is a specific form of necrotizing fasciitis and is located in the external genital organs and perianal region, causing thrombosis in the arteries feeding this region, gangrene in the skin and subcutaneous tissues, sepsis, and multiorgan failure.

The prognosis of Fournier's gangrene is closely related to the time of initiation of treatment. In cases where treatment is delayed, high mortality can be observed due to septic shock and related complications.

In laboratory tests, leukocytosis or leukopenia, anemia, and lymphopenia can be observed. In a study evaluating conditions that increase mortality with soft tissue necrosis, it was reported that high body mass index, abnormal leukocytes, CRP and platelet values were proportional to the severity of the disease.

Perianal abscess is a surgical emergency that is observed much more frequently than necrotizing fasciitis. Patients usually present with an erythematous swelling near the anus and hesitate to be examined. About 90% of idiopathic perianal abscesses occur due to infection of the cryptoglandular glands.

Although Fournier's gangrene has many different etiologies, it rarely occurs due to the progression of perianal abscess, and although it is difficult to distinguish between these two diseases in the diagnosis, the two diseases manifest themselves as different entities. In a study, higher IL17 levels were found in perianal abscess patients compared to the control group. Apart from this, we did not find any study on blood cytokine levels in patients with perianal abscess or Fournier's gangrene in our literature review.

In this study, blood cytokine levels will be evaluated in patients with Fournier's gangrene and perianal abscess, and the role of blood cytokine levels in the differential diagnosis of these two diseases will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients applying to the emergency department with Fournier's gangrene and perianal abscess.

Exclusion Criteria:

* Patients with primary immunodeficiency
* Crohn's patients
* HIV patients,
* Cancer patients,
* Pregnancy,
* Patients younger than 18 years and older than 88 years
* Patients who did not agree to participate in the study

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, patients who applied to the emergency department with rectal pain and were diagnosed with perianal abscess or Fournier's gangrene and volunteers in the same age range without any disease will be included.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Cytokines | 1 day
  Values in pg/ml of IL-1β, IFN-α2, IFN-γ, TNF-α, MCP-1 (CCL2), IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, IL-33

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Gaziosmanpasa Training and Research Hospital, Istanbul
  - Seyrantepe Hamidiye Etfal Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Diab J, Bannan A, Pollitt T. Necrotising fasciitis. BMJ. 2020 Apr 27;369:m1428. doi: 10.1136/bmj.m1428. No abstract available. PMID 32341079
- [Background] Wang JP, Cai C, Du JL, Shi HQ, Liu QW, Dai ZH, Zhong ZF. Role of interleukin-17 in the pathogenesis of perianal abscess and anal fistula: a clinical study on 50 patients with perianal abscess. ANZ J Surg. 2019 Mar;89(3):244-247. doi: 10.1111/ans.14874. Epub 2018 Oct 25. PMID 30362208
- [Background] Park SJ, Kim DH, Choi CI, Yun SP, Kim JH, Seo HI, Jo HJ, Jun TY. Necrotizing soft tissue infection: analysis of the factors related to mortality in 30 cases of a single institution for 5 years. Ann Surg Treat Res. 2016 Jul;91(1):45-50. doi: 10.4174/astr.2016.91.1.45. Epub 2016 Jun 30. PMID 27433464